CLINICAL TRIAL: NCT06580002
Title: Repurposing Riluzole for Augmenting Brain-Derived Neuropathic Factor (BDNF) Levels and Cognitive Function in Patients Experiencing Cancer-Related Cognitive Impairment: An Interventional Pilot Clinical Trial
Brief Title: Repurposing Riluzole for Cancer-Related Cognitive Impairment: A Pilot Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Alexandre Chan, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4994; UCI 24-05 (Other: UCI CFCCC)
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Sarcoma; Gastric Cancer; Lung Cancer; Head and Neck Cancer; Colorectal Cancer; Ovarian Cancer; Liver Cancer; Genitourinary Cancer; Gynecologic Cancer
MeSH Terms: conditions — Breast Neoplasms; Sarcoma; Stomach Neoplasms; Lung Neoplasms; Head and Neck Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Liver Neoplasms; Urogenital Neoplasms | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Riluzole (Experimental): Study participants randomized to this arm will take 50 mg of riluzole twice daily (every 12 hours) for 8 weeks
  Interventions: Drug: Riluzole
- Placebo (Placebo Comparator): Study participants randomized to this arm will take a placebo, that matches the appearance of 50 mg capsule of riluzole, twice daily (every 12 hours) for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riluzole — Given PO
  Other Names: RILUTEK
  Arms: Riluzole
Drug: Placebo — Given PO
  Arms: Placebo

SUMMARY:
This is a phase 2a, randomized, double-blinded, placebo-controlled pilot clinical trial determining the impact of riluzole therapy on circulating brain derived neuropathic factor (BDNF) levels of cancer survivors with cancer related cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients diagnosed with one of the following:

  1. Breast cancer exposed to treatment including chemotherapy, radiotherapy, surgery and/or other breast cancer interventions
  2. Non-breast cancer patients exposed to anthracyclines- or platinum-containing chemotherapy within the past 3 years
  3. Non-breast cancer patients exposed to other anticancer therapies within the past 3 years
* Washout from investigational interventions is up to the discretion of the Investigator. Concurrent participation in another intervention is allowable if judged by the Principal Investigator that this would not be scientifically or medically incompatible with this study.
* ≥18 years of age
* Perceived by patient or investigator that cognitive function has worsened since cancer diagnosis and/or beginning of cancer treatment
* Able to provide informed consent.
* Literacy in English, Chinese, Korean, Vietnamese, or Spanish, to complete the questionnaires.
* Patients must agree to complete and be able to complete the questionnaires and computerized assessments used to measure functional outcomes.

Note: Patients who have visual impairment or have degenerative conditions (e.g. Parkinsons's disease, etc.) can participate if they cannot complete computerized assessments, as long as they can still complete the questionnaires with assistance.

Exclusion Criteria:

* Presence of brain metastasis
* Unwilling to undergo neuropsychological assessments necessary for the study.
* Women who are breastfeeding, pregnant or are planning to get pregnant during the study period. Women of child-bearing potential (WOCBP) must have a negative pregnancy test at screening if there is suspicion of pregnancy.

  a. Female patients who are considered not to be of childbearing potential must have a history of being postmenopausal (with a minimum of 1 year without menses), tubal ligation, or hysterectomy.
* History of suspected hypersensitivity to riluzole or to any of its excipients.
* Patients taking or planned to take medications/substances with potential drug-drug interactions: pixantrone, current smoker (defined as having smoked within the last month), abametapir, cannabis, capmatinib, lapatinib, methotrexate, and levoketoconazole.
* Hepatic impairment as indicated by: AST or ALT ≥ 3x upper limit normal (ULN)
* Have serious pre-existing medical conditions that, in the judgment of the investigator, would preclude participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in circulating Brain-Derived Neurotrophic Factor (BDNF) levels over time in cancer survivors experiencing cognitive impairment (CRCI) | 8 weeks
  Comparing mean plasma BDNF values at each patient visit point, including before the intervention, at the midpoint, and at the endpoint of the study.

SECONDARY OUTCOMES:
Cognitive Function Scores (FACT-Cog) | 8 weeks
  Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) scores, including both cumulative and perceived cognitive impairment scores. These scores will be compared between intervention and placebo groups over time, with mixed effects models used to evaluate changes.There are four other scoring subscales in FACT-Cog v3: perceived cognitive impairments (PCI; 18 items); perceived cognitive abilities (7 items); impact of perceived cognitive impairment on QOL (4 items); and comments from others on cognitive function (4 items). Both total and PCI scores will be calculated in this study. Total score is calculated by summing scores from all the items and ranges from 0-148, and higher scores represent better subjective cognitive functioning. Similarly, PCI score is calculated by summing responses of all relevant items and ranges from 0 to 72.
Cognitive Function Scores (CANTAB) | 8 weeks
  The study will assess the effects of riluzole on cognitive function using the Cambridge Neuropsychological Test Automated Battery (CANTAB) scores across five cognitive domains. These scores will be compared between intervention and placebo groups over time, with mixed effects models used to evaluate changes. Cognitive domains of response speed, learning and memory, working memory, multitasking, and sustained attention will be assessed with CANTAB®. Using International Cognition and Cancer Task Force (ICCTF criteria), overall cognitive impairment is defined as ≥ 2 standard deviations below normative mean on at least 1 cognitive test or ≥ 1.5 standard deviations below normative mean on 2 or more tests.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Chan, PharmD, MPH, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California Irvine, Orange, California, United States